CLINICAL TRIAL: NCT00002203
Title: A Randomized, Multicenter Study of Epivir 150 Mg Bid, Retrovir 200 Mg Tid and a Protease Inhibitor Vs 3TC 150 Mg/ZDV 300 Mg Fixed Dose Tablet Given Bid With a Protease Inhibitor in HIV-Infected Patients
Brief Title: A Study of Two Anti-HIV Drug Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 280A; NZTA4001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; CD4-CD8 Ratio; Lamivudine; Patient Compliance; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Patient Compliance | interventions — lamivudine, zidovudine drug combination; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of taking lamivudine (3TC) plus zidovudine (ZDV) plus a protease inhibitor (PI) with taking the 3TC/ZDV combination tablet (Combivir) plus a PI. This study also examines how well patients follow the dosing schedules for these drugs.

Doctors believe that taking Combivir plus a PI may be as effective as taking 3TC plus ZDV plus a PI.

DETAILED DESCRIPTION:
It is hypothesized that a fixed-dose 3TC/ZDV tablet given bid in combination with a protease inhibitor is clinically equivalent in its effect on plasma HIV-1 RNA level to a conventional regimen of 3TC, ZDV, and a protease inhibitor.

Patients are stratified according to their current protease inhibitor therapy and randomized to receive open-label therapy of 1 Combivir tablet bid (Arm II) or an equivalent dose of 3TC and ZDV (Arm I), plus their current protease inhibitor for 16 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection documented by a licensed antibody ELISA assay and confirmed by Western blot, positive HIV blood culture, positive HIV serum antigen, or plasma viremia.
* CD4+ cell count of at least 300 cells/mm3.
* HIV-1 RNA less than 10,000 copies/ml by Roche Amplicor PCR assay.
* CDC Category A or B Classification for HIV infection (no clinical diagnosis of AIDS).
* Compliance with dosing schedule and protocol evaluations.

Prior Medication:

Required:

* 3TC at 150 mg bid, ZDV at 600 mg/day (200 mg tid or 300 mg bid), plus a marketed protease inhibitor (ritonavir, saquinavir, indinavir, or nelfinavir) at its recommended dose for at least 10 weeks.

Allowed:

* Inhaled corticosteroids for the treatment of asthma.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malabsorption syndromes affecting drug absorption (e.g., Crohn's disease and chronic pancreatitis).
* Enrollment in other investigational protocols.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapeutic agents.
* Nonnucleoside reverse transcriptase inhibitors.
* Other investigational agents.

Concurrent Treatment:

Excluded:

Radiation therapy.

Prior Medication:

Excluded:

* Cytotoxic chemotherapeutic and immunomodulating agents such as systemic corticosteroids, IF-2, alpha-IFN, beta-IFN, or gamma-IFN (except for inhaled corticosteroids for the treatment of asthma) within 4 weeks of study entry.
* HIV immunotherapeutic vaccine within 3 months of study entry.

Prior Treatment:

Excluded:

Radiation therapy within 4 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Pacific Oaks Med Ctr, Beverly Hills, California
  - Tower Infectious Diseases / Med Associates Inc, Los Angeles, California
  - Univ of North Carolina Hosps, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Infectious Diseases Physicians Inc, Annandale, Virginia
  - Univ of Wisconsin School of Medicine, Madison, Wisconsin
- San Juan AIDS Program, Santurce, Puerto Rico